CLINICAL TRIAL: NCT01842061
Title: Everyday Activity Supports You (EASY) Pilot Study
Acronym: EASY-Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Maureen C. Ashe, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: H13-00518
Record Dates: First submitted 2013-04-17; First posted 2013-04-29 (Estimated); Results first posted 2021-10-14 (Actual); Last update posted 2021-10-14 (Actual); Status verified 2021-09

CONDITIONS: Lifestyle
Keywords: active living; retirement
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active Living Program (Experimental): Participants in the intervention group will receive a self-management program designed to reduce sedentary behaviour and increase physical activity. Specifically, they will be given an EASY Program Manual with strategies to break up sitting time during the day and increase utilitarian activity; this will include a section on how to set, monitor and maintain achievable goals. They will also be offered a pedometer program, group education sessions and encouraged to use public transport by providing free bus tickets.
  Interventions: Behavioral: Active Living Program
- Education (Active Comparator): Control group participants will be offered monthly drop-in sessions that target information on general health and well-being unrelated to physical activity.
  Interventions: Behavioral: Education

INTERVENTIONS:
Behavioral: Active Living Program
  Arms: Active Living Program
Behavioral: Education
  Arms: Education

SUMMARY:
The investigators propose a 6-month, parallel, single-blind randomized controlled trial (RCT) feasibility study of a self-management program to reduce sedentary time and increase physical activity (Sit Less to Move More) in women aged 55-70 years. The primary aim is to determine feasibility and acceptability of the intervention; and the secondary aim is to test the effect of the intervention on the primary health outcome, physical activity (mean daily step count by accelerometry) at 6 months. The investigators will also conduct an economic evaluation and a process evaluation to guide a future larger study and to inform a scaled-up implementation plan.

ELIGIBILITY:
Inclusion Criteria:

* Healthy community-dwelling women aged 55-70 years who (via self-report) are not currently engaging (or in the previous 3 months) in any strength training, or <30 minutes brisk walking or moderate exercise/week
* are able to climb stairs and walk 400 meters (e.g., do not have a mobility disability).

Exclusion Criteria:

* Participants who receive treatment for medical conditions that preclude participation in a walking program

Ages: 55 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2013-05; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maureen C Ashe, PhD, Principal Investigator — University of British Columbia
Locations (1):
- Centre for Hip Health and Mobility, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ashe MC, Winters M, Hoppmann CA, Dawes MG, Gardiner PA, Giangregorio LM, Madden KM, McAllister MM, Wong G, Puyat JH, Singer J, Sims-Gould J, McKay HA. "Not just another walking program": Everyday Activity Supports You (EASY) model-a randomized pilot study for a parallel randomized controlled trial. Pilot Feasibility Stud. 2015;1:4. doi: 10.1186/2055-5784-1-4. Epub 2015 Jan 12. PMID 27175291
- [Derived] Gray SM, Chen P, Fleig L, Gardiner PA, McAllister MM, Puyat JH, Sims-Gould J, McKay HA, Winters M, Ashe MC. Can a Lifestyle Intervention Increase Active Transportation in Women Aged 55-70 years? Secondary Outcomes From a Pilot Randomized Controlled Trial. J Phys Act Health. 2018 Jun 1;15(6):411-416. doi: 10.1123/jpah.2016-0348. Epub 2018 Mar 23. PMID 29570005

RESULTS

PARTICIPANT FLOW:
Groups:
- Active Living Program: Participants in the intervention group will receive a self-management program designed to reduce sedentary behaviour and increase physical activity. Specifically, they will be given an EASY Program Manual with strategies to break up sitting time during the day and increase utilitarian activity; this will include a section on how to set, monitor and maintain achievable goals. They will also be offered a pedometer program, group education sessions and encouraged to use public transport by providing free bus tickets.
  Active Living Program
- Education: Control group participants will be offered monthly drop-in sessions that target information on general health and well-being unrelated to physical activity.
  Education
Period: Overall Study
Arm/Group | Active Living Program | Education
Started | 13 | 12
Completed | 12 | 8
Not Completed | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Living Program | Education | Total
Number analyzed (Participants) | 13 | 12 | 25
Age, Customized [Count of Participants; unit: Participants]
  aged 55-70 years | 13 | 12 | 25
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 1 participant in the intervention group did not complete the study, and 4 participants in the control group did not complete the study.
  Participants
    number analyzed (Participants) | 12 | 8 | 20
    Female | 12 | 8 | 20
    Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants] — Population: 1 participant from the intervention and 4 participants in the control group did not complete the study.
  participants
    Canada: number analyzed (Participants) | 12 | 8 | 20
    Canada | 12 | 8 | 20

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Study Recruitment and Retention
Description: The number of study participants recruited and finish the 6 month study (and final assessment).
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Active Living Program | Education
Number analyzed (Participants) | 12 | 8
Participants | 12 | 8

2. Secondary Outcome: Sedentary Time (Measured by Average Daily Percent)
Description: sedentary time (measured by average daily percent) as measured by accelerometry
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: percentage of day
Arm/Group | Active Living Program | Education
Number analyzed (Participants) | 12 | 7
percentage of day | 66.17 (7.06) | 67.23 (4.68)

3. Secondary Outcome: Physical Activity
Description: steps counts as measured by accelerometry
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: steps/day
Arm/Group | Active Living Program | Education
Number analyzed (Participants) | 12 | 7
steps/day | 7606 (3917) | 4593 (663)

4. Secondary Outcome: Body Composition
Description: body weight measured in kilograms
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: kgs
Arm/Group | Active Living Program | Education
Number analyzed (Participants) | 12 | 8
kgs | 67.33 (18.57) | 91.6 (19.04)

5. Secondary Outcome: Active Transportation
Description: Self reported description of minutes/week of active transportation (e.g., walking, cycling, etc.)
Time Frame: 6 months
Measure: Median (Inter-Quartile Range); unit: mins/week
Arm/Group | Active Living Program | Education
Number analyzed (Participants) | 12 | 8
mins/week | 396 [231 to 841.5] | 272.3 [0 to 321.8]

ADVERSE EVENTS:
Arm/Group | Active Living Program | Education
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/12
Other Adverse Events (participants affected / at risk) | 0/13 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No